CLINICAL TRIAL: NCT03242343
Title: A Multi-center Prospective Study to Evaluate the Safety and Effectiveness of the VasQ External Support for Arteriovenous Fistula
Brief Title: VasQ External Support for Arteriovenous Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laminate Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD0121
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Arterio-Venous Fistula; ESRD; Steal Syndrome; Aneurysm; Renal Failure; Renal Disease; Diabetes Mellitus; Kidney Failure
MeSH Terms: conditions — Arteriovenous Fistula; Kidney Failure, Chronic; Aneurysm; Renal Insufficiency; Kidney Diseases; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- VasQ device implantation (Experimental): Main study cohort: Prospective, multi-center, single-arm, open label, enrolling patients referred to surgical creation of new brachiocephalic fistula (BCF). The VasQ will be applied to the AV fistula in all patients. The primary effectiveness endpoint for this trial will be measured at 6 months and compared to a performance goal (PG). Safety will compare descriptively between AE rates for Steal, Infection, Aneurysm and Seroma. Patients will be followed up for an additional 18 months for a total of 2 years. Additionally, this trial has several secondary endpoints.
  Supplementary study cohort: 15 patients will be prospectively enrolled which are referred to surgical creation of a new forearm arteriovenous fistula. VasQ will be applied to the AV fistula in all patients. Patients will be followed in the same manner as in the Main study cohort, however, the data will be reported separately and not be part of the analysis sets for the study primary and secondary endpoints.
  Interventions: Device: VasQ

INTERVENTIONS:
Device: VasQ — An external support device for AV fistula

SUMMARY:
This is a prospective clinical study of the VasQ external support for arteriovenous fistulas. The device is designed to improve fistula outcomes by optimizing the geometrical configuration of the fistula, influencing hemodynamics, minimizing turbulence and promote laminar flow.

All patients will be implanted with the VasQ device and will be followed up for a duration of 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Main study cohort: Patients referred for creation of a new brachiocephalic fistula who consent to take part in the study and which are not indicated for a more distal fistula per treatment guidelines.

   Supplementary study cohort: Patients referred for creation of a new forearm fistula who consent to take part in the study.
2. Male and female participants.
3. Age 18-80 years.
4. Patients willing and able to attend follow up visits over a period of 24 months.

Exclusion Criteria:

1. Patients with the planned index procedure being a revision surgery of an existing fistula.
2. Main study cohort: Target artery smaller than 2.5 mm or larger than 6 mm in inner diameter by preoperative ultrasound.

   Supplementary study cohort: Target artery smaller than 2 mm or larger than 4.1 mm in inner diameter by preoperative ultrasound.
3. Main study cohort: Target vein smaller than 2.5 mm in inner diameter by preoperative ultrasound.

   Supplementary study cohort: Target vein smaller than 2 mm in inner diameter by preoperative ultrasound.
4. Significantly stenotic target vein on the side of surgery (≥50%) as diagnosed on preoperative ultrasound. (Scan should include the area between the planned anastomosis site and the Axillary vein.)
5. Unusual anatomy or vessel dimensions (observed on pre-operative ultrasound or intraoperatively) and which preclude adequate fit of the VasQ.
6. Patients with central venous stenosis or obstruction on the side of surgery.
7. Depth of vein greater than 8 mm (on ultrasound) on side of surgery.
8. Known coagulation disorder.
9. Congestive heart failure NYHA class ≥ 3.
10. Prior steal on the side of surgery.
11. Known allergy to nitinol.
12. Life expectancy less than 30 months.
13. Patients expecting to undergo kidney transplant within 6 months of enrollment.
14. Women of child bearing age without documented current negative pregnancy test.
15. Inability to give consent and/or comply with the study follow up schedule.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2022-04-03 (Actual)

PRIMARY OUTCOMES:
Primary Patency of AVF | 6 months post AVF creation
  Proportion of patients with freedom from intervention since device placement
Occurrence of safety events | Device implantation to 6 months post AVF creation
  The occurrence per patient access related safety events

CONTACTS AND LOCATIONS:
Overall Officials: Noam Zilberman, Study Director — Laminate Medical Technologies Ltd.
Locations (15):
- United States (15):
  - Grandview Medical Center, Birmingham, Alabama
  - Arizona Kidney Disease & Hypertension Center, Phoenix, Arizona
  - Saint Francis Medical Center, Peoria, Illinois
  - Lutheran Medical Group/Indiana Ohio Heart, Fort Wayne, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Albany Medical College, Albany, New York
  - Montefiore Medical Center, New York, New York
  - Charlotte PA, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Wexner Meidcal Center, Columbus, Ohio
  - Greenville Health System, Greenville, South Carolina
  - Cardiothoracic and Vascular Surgeons, P.A., Austin, Texas
  - Methodist DeBakey Heart and Vascular Center,The Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chemla E, Velazquez CC, D'Abate F, Ramachandran V, Maytham G. Arteriovenous fistula construction with the VasQ external support device: a pilot study. J Vasc Access. 2016 May 7;17(3):243-8. doi: 10.5301/jva.5000527. Epub 2016 Apr 14. PMID 27079670
- See also: Related Info — http://www.laminatemedical.com/